CLINICAL TRIAL: NCT02291653
Title: Comparing the Novel McGrath MAC EMS Videolaryngoscope With Conventional Direct Laryngoscopy During Child Resuscitation: a Randomized Crossover Mannequin Study of Paramedic Students
Brief Title: Pediatric Endotracheal Intubation
Acronym: EMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: International Institute of Rescue Research and Education (Other)
Responsible Party: Principal Investigator, Lukasz Szarpak, Lukasz Szarpak, National Institute of Cardiology, Warsaw, Poland
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ETI/2014/17
Record Dates: First submitted 2014-11-11; First posted 2014-11-14 (Estimated); Last update posted 2014-12-05 (Estimated); Status verified 2014-12

CONDITIONS: Cardiac Arrest; Intubation, Endotracheal
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intubation without chest compressions (Experimental): Endotracheal intubation of pediatric mannikin during resuscitation without chest compressions.
  Interventions: Device: McGrath; Device: MIL
- Intubation with uninterrupted chest compressions (Experimental): Endotracheal intubation of pediatric mannikin during resuscitation with uninterrupted chest compressions. In order to simulate the difficulties associated with intubation during uninterrupted chest compressions, CPR was performed by using LUCAS-2 (Physio-Control, Redmond, WA, U.S.).
  Interventions: Device: McGrath; Device: MIL

INTERVENTIONS:
Device: McGrath — video-laryngoscopy
  Other Names: McGrath MAC EMS
Device: MIL — direct-laryngoscopy
  Other Names: Miller Laryngoscope

SUMMARY:
We hypothesized that the McGrath MAC EMS is beneficial for intubation of pediatric manikins while performing CPR. In the current study, we compared effectiveness of the McGrath MAC EMS and MIL laryngoscopes in child resuscitation with and without CC.

ELIGIBILITY:
Inclusion Criteria:

* Give voluntary consent to participate in the study
* paramedic student

Exclusion Criteria:

* Not meet the above criteria
* Wrist or Low back diseases

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2014-11; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Success of intubation | 1 day
  effectiveness of first, second and third intubation attempts and overall effectiveness of intubation by participants

SECONDARY OUTCOMES:
Intubation time | 1 day
  time in seconds required for a successful intubation attempt
Cormack-Lehane grading | 1 day
  self-reported percentage the vocal cord visualization using the Cormack-Lehane grading (grade 1-4)

CONTACTS AND LOCATIONS:
Overall Officials: Lukasz Szarpak, Principal Investigator — Institute of Cardiology
Locations (1):
- International Institute of Rescue Research and Education, Warsaw, Masovia, Poland